CLINICAL TRIAL: NCT03793660
Title: Safety and Efficacy of Biotherapy in Rheumatoid Aarthritis and Spondyloarthritis. A Clinical Multicentric Study: Biologic National Registry (BINAR)
Brief Title: Biologic National Registry
Acronym: BINAR
Status: Completed | Type: Observational
Sponsor: Dacima Consulting (Other)
Collaborators: Ligue Tunisienne Anti Rhumatismale (Unknown)
Responsible Party: Sponsor
Other Study IDs: DAC-004-LITAR
Record Dates: First submitted 2018-12-29; First posted 2019-01-04 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Arthritis, Rheumatoid; Spondylitis
Keywords: Biologic; Safety; LITAR; DACIMA; Tunisia
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
BINAR is an open and multicentric Tunisian national registry performed by nearly 100 rheumatologists

DETAILED DESCRIPTION:
BINAR is a Tunisian, descriptive, non-interventional, multicenter and prospective clinical study performed in rheumatology consultations, of both public and liberal sectors. Eligible patients are recruited by successive inclusions until the end of the recruitment period, set at one year. A Scientific Committee validates the scientific writing, a Steering Committee supervises the clinical operations of the project and a Data Review Committee supervises the management of the data and carries out all the missions of audit and control of validity of the collected data, as well as the planning of statistical analysis.

Collected data are managed by the DACIMA Clinical Suite®, the electronic data capture platform which complies with the FDA 21 CFR part 11 requirements (Food and Drug Administration 21 Code of Federal Regulations part 11), the HIPAA specifications (Health Insurance Portability and Accountability Act), and the ICH standards (International Conference on Harmonisation).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient followed for rheumatoid arthritis according to ACR EULAR criteria or spondylitis including all disorders (axial, peripheral, enthesitis).
* Patient on biological treatment at the time of inclusion
* First biological treatment initiated ≤ 2 years
* Informed consent, read and signed

Exclusion Criteria:

* Evolutionary neoplasia at the time of inclusion
* Other associated systemic diseases, except Sjögren's Syndrome
* Consent not obtained
* Pregnant or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated with biologic for rheumatoid arthritis or spondylitis
Sampling Method: Non-Probability Sample
Enrollment: 439 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Safety assessment of biotherapy - Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]: Occurrence of infection or tuberculosis or death or neoplasia or any other treatment-related side effect of biotherapy | Up to two years of follow-up
  Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] : occurrence of infection or tuberculosis or death or neoplasia or any other treatment-related side effect of biotherapy

SECONDARY OUTCOMES:
Assessment of Rheumatoid Arthritis Activity | At baseline and at two years follow-up
  Number of patients with disease Activity Score (DAS) < 2.6
Health Assessment Questionnaire | At baseline
  HAQ assessment for Rheumatoid Arthritis patients (range score 0-3)
Assessment of Spondylitis Fonctional Activity | At baseline and at two years follow-up
  Bath Ankylosing Spondylitis Fonctional Index measurement (BASFI) : (range score 0-10)
Assessment of Spondylitis Disease Activity | At baseline and at two years follow-up
  Bath Ankylosing Spondylitis Disease Activity Index measurement (BASDAI) : (range score 0-10)
Assessment of Spondylitis Activity | At baseline and at two years follow-up
  Number of patients with Ankylosing Spondylitis Disease Activity Score (ASDAS) < 2.1

CONTACTS AND LOCATIONS:
Overall Officials: Samir Kochbati, MD, Study Chair — LITAR : Ligue Tunisienne Anti Rhumatismale; Kawther Ben Abdelghani, MD, Principal Investigator — LITAR : Ligue Tunisienne Anti Rhumatismale
Locations (10):
- Tunisia (10):
  - Rheumatology Department - Habib Thameur, Ben Arous
  - Rheumatology Department - HMPIT, Ben Arous
  - Rheumatology Department - Tahar Sfar, Mahdia
  - Rheumatology Department - Institut Mohamed Kassab d'Orthopédie, Manouba
  - Rheumatology Department - Fattouma Bourguiba, Monastir
  - Rheumatology Department - Hédi Chaker, Sfax
  - Rheumatology Department - Farhat Hached, Sousse
  - Rheumatology Department - Charles Nicolle, Tunis
  - Rheumatology Department - La Rabta, Tunis
  - Rheumatology Department - Mongi Slim, Tunis

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Social Media Group of the Project — https://www.facebook.com/groups/1611044669000801/about/